CLINICAL TRIAL: NCT02538835
Title: The Effect of Group Treatment for Depression: A Randomised Controlled Study of Metacognitive Therapy, Mindfulness and Support Groups
Brief Title: The Effect of Group Treatment for Depression: A Study of Metacognitive Therapy, Mindfulness and Support Groups
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Center for Kognitive Terapier og Supervision (Unknown)
Responsible Party: Principal Investigator, Tonny Elmose Andersen, phd., Associate Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46332
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy; Population Groups; Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Metacognitive Therapy (Experimental)
  Interventions: Behavioral: Metacognitive therapy
- Mindfulness based cognitive therapy (Active Comparator)
  Interventions: Behavioral: Mindfulness based cognitive therapy, group
- Support groups (Placebo Comparator)
  Interventions: Behavioral: Support groups

INTERVENTIONS:
Behavioral: Metacognitive therapy — Group format, 10-12 participants in each group. 8 weekly sessions of two hours each.
  Arms: Metacognitive Therapy
Behavioral: Mindfulness based cognitive therapy, group — Group format, 10-12 participants in each group. 8 weekly sessions of two hours each following the manual described by Williams, Zindel & Segal.
  Arms: Mindfulness based cognitive therapy
Behavioral: Support groups — Group format, 10-12 participants in each group. The sessions will only be of supportive character and will not focus on changing or restructuring thoughts, scripts or thought patterns. The format will follow a manual but compared to the other intervention groups the format allow participants to suggests themes for discussions.
  Arms: Support groups

SUMMARY:
This study evaluates the effect of metacognitive group therapy on depression compared to mindfulness groups and supportive groups. The participants, all with a history of depression and with current symptoms of depression, will be randomized to one of the three group interventions.

DETAILED DESCRIPTION:
Metacognitive therapy (MCT) show promising results in alleviating depressive symptoms and reducing relapse of depression. However studies of MCT as a group intervention is limited and higher quality studies of the effectiveness of MCT is warranted. The present study aim to produce more conclusive evidence on the effect of MCT comparing MCT in groups with both and active control group and mindfulness based cognitive therapy (MBCT), which together with pharmacotherapy is currently one of the preferred treatment choices. Currently pharmacotherapy, cognitive therapy and MBCT seem to help 40-58% of the patients efficiently. The current studies of MCT indicate that this intervention may help a higher proportion of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate
* History of clinical depression
* Current depressive symptoms
* Verbal and cognitive abilities to complete the questionnaires during the study
* Stable medication - if any medication is ordinated
* Speaks fluently danish

Exclusion Criteria:

* If criteria for psychosis, bipolar disorder or personality disorder is matched
* known brain damage or mental retardation
* substance abuse
* women who are pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2018-08; Primary Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on Hamilton depression scale | 8 weeks
Change from baseline on Hamilton depression scale | 32 weeks

SECONDARY OUTCOMES:
Change from baseline on Becks depression inventory | 8 weeks
Change from baseline on Becks depression inventory | 32 weeks
Change from baseline on Becks Anxiety Inventory | 8 weeks
Change from baseline on Becks Anxiety Inventory | 32 weeks
Change from baseline on Ruminative Response Scale | 8 weeks
Change from baseline on Ruminative Response Scale | 32 weeks
Change from baseline on Metacognitive questionnaire | 8 weeks
Change from baseline on Metacognitive questionnaire | 32 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Odense, Southern Denmark, Denmark